CLINICAL TRIAL: NCT03870399
Title: Phase II Study of Hormone Therapy With Tamoxifen in Patients With Well Differentiated Neuroendocrine Tumors and Hormone Receptor Positive Expression
Brief Title: Study of Tamoxifen in Well Differentiated Neuroendocrine Tumors and Hormone Receptor Positive Expression
Acronym: HORMONET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AC Camargo Cancer Center (Other)
Collaborators: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Principal Investigator, Rachel Riechelmann, Head of Clinical Oncology Department, AC Camargo Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2626/18; NCT04123262 (obsolete NCT alias)
Record Dates: First submitted 2019-03-06; First posted 2019-03-12 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Neuroendocrine Tumors; Progesterone Receptor Positive Tumor; Estrogen Receptor Positive Tumor
Keywords: neuroendocrine tumor; tamoxifen; Progesterone Receptor; Estrogen Receptor
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Tamoxifen

STUDY DESIGN:
Intervention Model Description: A single-arm, unicentric, single-stage clinical study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tamoxifen (Experimental): The participants will receive tamoxifen 20mg orally once daily with a glass of water. Each cycle will be defined for 42 days (6 weeks).
  Interventions: Drug: Tamoxifen

INTERVENTIONS:
Drug: Tamoxifen — The treatment to be used will be tamoxifen 20mg orally once daily.

SUMMARY:
This is a single-arm, unicentric, single-stage clinical study of tamoxifen for patients with well differentiated neuroendocrine tumors and radiological progression with positive (> 1 percent) HR (estrogen and / or progesterone) expression by IHC. It will evaluate if Tamoxifen exerts antitumor action in patients with well differentiated NET and positive for the expression of HR, estrogen and / or progesterone.

DETAILED DESCRIPTION:
Neuroendocrine tumors (NET) are rare neoplasms, but with increasing incidence and prevalence in the last decades. Although they may manifest in the most diverse tissues, the vast majority of cases will affect organs of the digestive tract and lung. At diagnosis, more than half of the cases present metastatic disease, and among patients with localized disease, up to one-third will have recurrence of the disease. Unfortunately, the minority of patients with metastatic disease are eligible for curative intent. Although there are many types of NET, they are often studied together as a group because their cells share common histological findings, have special secretory granules, and the ability to secrete bioactive amines and polypeptide hormones. Approximately 25 percent of the tumors present functional hormonal syndromes (situation of great morbidity for these patients), being the carcinoid syndrome, the most common one. From the molecular point of view, these neoplasias are largely dependent on the activation of the mTOR pathway and neoangiogenesis. Another striking feature of neuroendocrine cells is the expression of cell surface hormone receptors whose activation or blockade may exert an important regulatory function. The discovery of somatostatin, and consequently its receptors, is one of the major advances in the treatment of this neoplasm. Due to the increased ability of somatostatin to inhibit the secretion of several hormones, its antitumor property has long been studied. However, only after the development of synthetic long-life formulations can their use be used in clinical practice. Well-differentiated neuroendocrine tumors (G1 and G2 according to World Health Organization (WHO) classification) present in more than 80 percent of somatostatin receptor cases. In this population, the use of somatostatin analogues promotes symptomatic improvement of functioning syndromes in the order of 70 to 77 percent and biochemical improvement around 50 percent . Regarding antiproliferative activity, two phase III studies evaluated the role of octreotide LAR and of lanreotide autogel, both somatostatin analogs, in the population of well differentiated tumors and, almost entirely, somatostatin receptor hyperexpressors when evaluated by octreoscan. In these studies, the use of somatostatin analogue was associated with reduced risk of progression or death from 53 percent to 66 percent when compared to placebo. Currently, this class of drugs is often considered as the first treatment option for patients with progressing metastatic disease, when the strategy of watchful waiting is not opted for (because they are tumors of sometimes indolent behavior, some cases are selected for observation only). In general, there are few options for systemic therapies that are approved for these tumors in addition to somatostatin analogs (mTOR and antiangiogenic inhibitors), none of which clearly demonstrate overall survival gain, are costly and none are available for use in the public health system (SUS). Therefore, it is very important to develop studies with new therapies for patients with NET, especially, molecularly defined therapies with greater access to patients. In this context, other anti-hormonal therapies could be explored in patients with NET, such as the role of the sex hormones estrogen and progesterone, as well as their receptors. A few studies have evaluated the expression of estrogen and progesterone receptors in NET and suggest interesting results. One of the largest series was conducted at the AC Camargo Cancer Center where the immunohistochemical expression of these receptors was evaluated in 96 patients with NET from various sites. About 35 percent of the cases presented positivity for some hormonal receptor (HR) in the tumor tissue. Among the HR positive cases, there was no difference between sex, more frequent in thin, pancreatic and lung tumors and in well differentiated tumors (G1 and G2 by the WHO). Viale et al. Evaluated the expression of progesterone receptors (PR) in 96 patients with pancreatic neuroendocrine tumors. Nuclear immunoreactivity for PR was observed in 58 percent of cases, with no difference in PR expression according to gender, age, or functioning syndromes. About 163 primary tumors of the gastroenteropancreatic site and 115 metastases were evaluated by Zimmermann and colleagues for expression of female hormone receptors. Progesterone receptor was more frequently found in pancreatic tumors and rarely in non-pancreatic (p <0.001), estrogen receptor was more frequently expressed in non-pancreatic tumors (<0.001) and in women (p: 0.019). There was no difference between primary site and presence of metastases. Apparently, HR positive tumors may present a more favorable evolution. A study evaluated 160 patients with pancreatic neuroendocrine tumors operated for expression by PTEN immunohistochemistry (negative regulator of the mTOR pathway) and PR. Approximately 69 percent of the cases were positive for PR and PTEN, 28 percent were positive for one of the two markers and only 3 percent were negative for both. Combined positivity for PTEN and PR was associated with metastasis-free survival in stages I and II (p <0.001) and overall survival in all patients (p <0.001), even after adjustment for other prognostic variables. Patients with negative PR and PTEN tumors had the shorter survival times when compared to those who had only one or both markers (p <0.001). 9 Similarly, other author demonstrated a retrospective analysis of 277 patients with neuroendocrine tumors (95 percent vs. 76 percent, p <0.05), and a higher survival rate (p <0.05) than in the control group (p <0.05) 0.015). Even rarer in the literature is the role of antiestrogen therapies as a form of control of this neoplasia. Case reports point to antiproliferative activity of tamoxifen in patients with NET and, in some cases, patients presenting more than 12 months of disease control.11 Reports of control of carcinoid syndrome and even regression of associated retroperitoneal fibrosis have also been described. However, the only study to assess the activity of tamoxifen in neuroendocrine tumors dates back to 1984. Sixteen patients were evaluated clinical benefit in only 19 percent of cases and no radiological response. However, in this study, no patient was previously selected for HR tumor expression or degree of differentiation, which the investigators believe limited benefit in disease control. Therefore, based on the premise that there is a need for research and treatment strategies for this rare neoplasm; there is clear therapeutic embezzlement in the public heath system due to the high cost of the treatments approved in the country for this neoplasia; NET are tumors that may present positivity to estrogen and / or progesterone receptors; evidence points to the possibility of antiproliferative effect using hormonal therapy, the investigators propose a phase II study of tamoxifen for patients with well differentiated NET and positive for HR, estrogen and / or progesterone expression.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Histological diagnosis of well differentiated NET (typical and atypical lung carcinoids, NET G1, NET G2 of all gastroenteropancreatic sites and pancreatic NET G3 according to WHO 2017 classification) 20 advanced / metastatic, inoperable, with no possibility of curative treatment
* Immunohistochemical expression ≥ 1 percent for estrogen and / or progesterone receptor
* Disease with radiological progression (at least 10 percent tumor volume growth) in the last 12 months before day 1 cycle 1.
* No possibility of established treatments due to lack of access, risk of toxicities or without clinical indication. Patients who meet criteria for watchful waiting (low-dose disease and non-functioning NET) may be included.
* Measurable disease
* ECOG performance scale 0 to 2.
* Adequate organic function as defined by the following criteria:

  * serum aspartate aminotransferase (AST), serum alanine aminotransferase (ALT) ≤ 2.5 times the upper limit of local laboratory normality (LSN-LL);
  * Total serum bilirubin ≤ 2.0 x ULN-LL;
  * Absolute neutrophil count ≥ 1,500 / mm^3;
  * Platelet count ≥ 80,000 / mm^3;
  * Hemoglobin ≥ 9.0 g / dL;
  * Estimated creatinine clearance by the MDRD equation ≥ 30ml / min
* Albumin ≥ 3.5 g / dL;
* INR ≤ 1.5
* Term of free and informed consent signed by the patient or legal representative.

Exclusion Criteria:

* Patients already on tamoxifen, but other prior treatment are allowed
* Patients with aggressive disease requiring cytotoxic therapy or locoregional therapies (eg hepatic embolization)
* A history of serious clinical or psychiatric illness that, by clinical judgment, may involve participation risk in this study
* Patients participating in other protocols with experimental drugs.
* Patients with oral food difficulties.
* Patients who underwent major recent surgery less than 4 weeks previously.
* Patients receiving chemotherapy or other oncologic therapy for less than 3 weeks.
* Patients who use oral anticoagulation
* Previous history of deep vein thrombosis or pulmonary embolism in the last 12 months.
* Pregnant or lactating patients.
* Patients with postmenopausal vaginal bleeding with no defined etiology.
* Patients with breast cancer who need to use tamoxifen for this neoplasm
* Another synchronous neoplasm that requires systemic treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2023-05-13 (Actual); Study Completion 2023-05-13 (Actual)

PRIMARY OUTCOMES:
Disease control rate | at 24 weeks after initiation of tamoxifen (at the end of cycle 6 - each cycle is 28 days)
  Defined by absence of radiological progression in conventional imaging examinations by RECIST 1.1. Isolated increase of biomarker (chromogranin A) or specific hormone will not be considered progression.

SECONDARY OUTCOMES:
Progression-free survival | Through study completion, an average of 5 years
  Defined by time from tamoxifen day 1 cycle 1 to death from any cause or radiological progression by RECIST 1.1, whichever occurs first. Patients alive and without progression at the time of study analysis will be censored for time-to-event analysis.
Rate of Biochemical response | Through study completion, an average of 5 years
  Defined by at least 30 percent drop in the marker (chromogranin and / or specific hormone) at any time of treatment in relation to pre-treatment value
Radiological response rate | Through study completion, an average of 5 years
  Assessed by RECIST criteria 1.1
Disease control rate | Through study completion, an average of 5 years
  defined by absence of radiological progression by RECIST 1.1 criteria, according to the intensity of expression by immunohistochemistry (IHC) of HR and also according to primary site (pancreas, gastrointestinal or lung)
Incidence of Treatment-related Adverse Events | Through study completion, an average of 5 years
  Frequency of adverse events of grades 2 or more by Common Adverse Event Toxicity Criteria (CTCAE) version 5.0

OTHER OUTCOMES:
PET-CT gallium-68 intake variation | Through study completion, an average of 3 years
  Evaluate possible variations in intensity of intake between PET-CT gallium-68 pre-treatment and 12 weeks after initiation of tamoxifen as a continuous variable for each capture lesion.
PET-CT gallium-68 number variation | Through study completion, an average of 3 years
  Evaluate possible variations in number of sites with intake between PET-CT gallium-68 pre-treatment and 12 weeks after initiation of tamoxifen as a continuous variable for each capture lesion.
CTC positivity rate | Through study completion, an average of 3 years
  Evaluate the percentage of CTC positivity in NET.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel SP Riechelmann, Phd, Principal Investigator — Fundacao Antonio Prudente; Jonathan R Strosberg, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (2):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States
- AC Camargo Cancer Center, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yao JC, Hassan M, Phan A, Dagohoy C, Leary C, Mares JE, Abdalla EK, Fleming JB, Vauthey JN, Rashid A, Evans DB. One hundred years after "carcinoid": epidemiology of and prognostic factors for neuroendocrine tumors in 35,825 cases in the United States. J Clin Oncol. 2008 Jun 20;26(18):3063-72. doi: 10.1200/JCO.2007.15.4377. PMID 18565894
- [Background] Caplin ME, Buscombe JR, Hilson AJ, Jones AL, Watkinson AF, Burroughs AK. Carcinoid tumour. Lancet. 1998 Sep 5;352(9130):799-805. doi: 10.1016/S0140-6736(98)02286-7. PMID 9737302
- [Background] Modlin IM, Pavel M, Kidd M, Gustafsson BI. Review article: somatostatin analogues in the treatment of gastroenteropancreatic neuroendocrine (carcinoid) tumours. Aliment Pharmacol Ther. 2010 Jan 15;31(2):169-88. doi: 10.1111/j.1365-2036.2009.04174.x. Epub 2009 Oct 21. PMID 19845567
- [Background] Caplin ME, Pavel M, Ruszniewski P. Lanreotide in metastatic enteropancreatic neuroendocrine tumors. N Engl J Med. 2014 Oct 16;371(16):1556-7. doi: 10.1056/NEJMc1409757. No abstract available. PMID 25317881
- [Background] Rinke A, Muller HH, Schade-Brittinger C, Klose KJ, Barth P, Wied M, Mayer C, Aminossadati B, Pape UF, Blaker M, Harder J, Arnold C, Gress T, Arnold R; PROMID Study Group. Placebo-controlled, double-blind, prospective, randomized study on the effect of octreotide LAR in the control of tumor growth in patients with metastatic neuroendocrine midgut tumors: a report from the PROMID Study Group. J Clin Oncol. 2009 Oct 1;27(28):4656-63. doi: 10.1200/JCO.2009.22.8510. Epub 2009 Aug 24. PMID 19704057
- [Background] Viale G, Doglioni C, Gambacorta M, Zamboni G, Coggi G, Bordi C. Progesterone receptor immunoreactivity in pancreatic endocrine tumors. An immunocytochemical study of 156 neuroendocrine tumors of the pancreas, gastrointestinal and respiratory tracts, and skin. Cancer. 1992 Nov 1;70(9):2268-77. doi: 10.1002/1097-0142(19921101)70:93.0.co;2-x. PMID 1356613
- [Background] Zimmermann N, Lazar-Karsten P, Keck T, Billmann F, Schmid S, Brabant G, Thorns C. Expression Pattern of CDX2, Estrogen and Progesterone Receptors in Primary Gastroenteropancreatic Neuroendocrine Tumors and Metastases. Anticancer Res. 2016 Mar;36(3):921-4. PMID 26976979
- [Background] Estrella JS, Broaddus RR, Mathews A, Milton DR, Yao JC, Wang H, Rashid A. Progesterone receptor and PTEN expression predict survival in patients with low- and intermediate-grade pancreatic neuroendocrine tumors. Arch Pathol Lab Med. 2014 Aug;138(8):1027-36. doi: 10.5858/arpa.2013-0195-OA. PMID 25076292
- [Background] Kim SJ, An S, Lee JH, Kim JY, Song KB, Hwang DW, Kim SC, Yu E, Hong SM. Loss of Progesterone Receptor Expression Is an Early Tumorigenesis Event Associated with Tumor Progression and Shorter Survival in Pancreatic Neuroendocrine Tumor Patients. J Pathol Transl Med. 2017 Jul;51(4):388-395. doi: 10.4132/jptm.2017.03.19. Epub 2017 Jun 8. PMID 28597868
- [Background] Arganini M, Spinelli C, Cecchini GM, Miccoli P. Long term treatment with tamoxifen for metastatic carcinoid tumor. Acta Chir Belg. 1989 Jul-Aug;89(4):209-11. PMID 2800857
- [Background] Myers CF, Ershler WB, Tannenbaum MA, Barth R. Tamoxifen and carcinoid tumor. Ann Intern Med. 1982 Mar;96(3):383. doi: 10.7326/0003-4819-96-3-383_1. No abstract available. PMID 7059114
- [Background] Biasco E, Antonuzzo A, Galli L, Baldi GG, Derosa L, Marconcini R, Farnesi A, Ricci S, Falcone A. Small-bowel neuroendocrine tumor and retroperitoneal fibrosis: efficacy of octreotide and tamoxifen. Tumori. 2015 Mar 20;101(1):e24-8. doi: 10.5301/tj.5000259. PMID 25702678
- [Background] Stathopoulos GP, Karvountzis GG, Yiotis J. Tamoxifen in carcinoid syndrome. N Engl J Med. 1981 Jul 2;305(1):52. doi: 10.1056/NEJM198107023050115. No abstract available. PMID 7231519
- [Background] Moertel CG, Engstrom PF, Schutt AJ. Tamoxifen therapy for metastatic carcinoid tumor: a negative study. Ann Intern Med. 1984 Apr;100(4):531-2. doi: 10.7326/0003-4819-100-4-531. No abstract available. PMID 6200021
- [Background] Harvey JM, Clark GM, Osborne CK, Allred DC. Estrogen receptor status by immunohistochemistry is superior to the ligand-binding assay for predicting response to adjuvant endocrine therapy in breast cancer. J Clin Oncol. 1999 May;17(5):1474-81. doi: 10.1200/JCO.1999.17.5.1474. PMID 10334533
- [Background] Goldhirsch A, Glick JH, Gelber RD, Coates AS, Thurlimann B, Senn HJ; Panel members. Meeting highlights: international expert consensus on the primary therapy of early breast cancer 2005. Ann Oncol. 2005 Oct;16(10):1569-83. doi: 10.1093/annonc/mdi326. Epub 2005 Sep 7. PMID 16148022
- [Background] Krebs MG, Hou JM, Sloane R, Lancashire L, Priest L, Nonaka D, Ward TH, Backen A, Clack G, Hughes A, Ranson M, Blackhall FH, Dive C. Analysis of circulating tumor cells in patients with non-small cell lung cancer using epithelial marker-dependent and -independent approaches. J Thorac Oncol. 2012 Feb;7(2):306-15. doi: 10.1097/JTO.0b013e31823c5c16. PMID 22173704
- [Background] Crippa S, Partelli S, Belfiori G, Palucci M, Muffatti F, Adamenko O, Cardinali L, Doglioni C, Zamboni G, Falconi M. Management of neuroendocrine carcinomas of the pancreas (WHO G3): A tailored approach between proliferation and morphology. World J Gastroenterol. 2016 Dec 7;22(45):9944-9953. doi: 10.3748/wjg.v22.i45.9944. PMID 28018101
- [Background] Furr BJ, Jordan VC. The pharmacology and clinical uses of tamoxifen. Pharmacol Ther. 1984;25(2):127-205. doi: 10.1016/0163-7258(84)90043-3. No abstract available. PMID 6438654
- [Background] Shiau AK, Barstad D, Loria PM, Cheng L, Kushner PJ, Agard DA, Greene GL. The structural basis of estrogen receptor/coactivator recognition and the antagonism of this interaction by tamoxifen. Cell. 1998 Dec 23;95(7):927-37. doi: 10.1016/s0092-8674(00)81717-1. PMID 9875847
- [Background] Yao JC, Shah MH, Ito T, Bohas CL, Wolin EM, Van Cutsem E, Hobday TJ, Okusaka T, Capdevila J, de Vries EG, Tomassetti P, Pavel ME, Hoosen S, Haas T, Lincy J, Lebwohl D, Oberg K; RAD001 in Advanced Neuroendocrine Tumors, Third Trial (RADIANT-3) Study Group. Everolimus for advanced pancreatic neuroendocrine tumors. N Engl J Med. 2011 Feb 10;364(6):514-23. doi: 10.1056/NEJMoa1009290. PMID 21306238
- [Derived] Barros MJ, Strosberg J, Al-Toubah T, de Jesus VHF, Durant L, Mello CA, Felismino TC, De Brot L, Taboada RG, Donadio MD, Riechelmann RP. HORMONET: a phase II trial of tamoxifen for estrogen/progesterone receptor-positive neuroendocrine tumors. Ther Adv Med Oncol. 2023 Jul 29;15:17588359231186041. doi: 10.1177/17588359231186041. eCollection 2023. PMID 37529158

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-03-06): https://cdn.clinicaltrials.gov/large-docs/99/NCT03870399/Prot_SAP_ICF_000.pdf